CLINICAL TRIAL: NCT05834205
Title: Effects of Plyometric Training Versus Bowling Drills on Agility and Speed Among Cricket Fast Bowlers
Brief Title: Effects of Plyometric Training Versus Bowling Drills on Fast Bowlers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/0401
Record Dates: First submitted 2023-04-18; First posted 2023-04-28 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-09

CONDITIONS: Sports Physical Therapy
Keywords: agility, cricket sport, drills, plyometric
MeSH Terms: interventions — Plyometric Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Plyometric Training (Experimental): Plyometric training regime:
  Ankle hops, jump squats, box jump, overhead medicine ball, plyometric push-up, rotational wall with 16x2 reps for week 1&2.
  Ankle hops, jump squats, box jump, overhead medicine ball, plyometric push-up, rotational wall with 10x3 reps for week 3&4.
  Ankle hops, jump squats, box jump, depth jump and alternate lunge jump, overhead medicine ball, plyometric push-up, rotational wall with 8x3 reps for week 5&6.
  Interventions: Other: Plyometric Training
- Drills (Active Comparator): Fast bowling drills (hitting a target, football throw, fast bowler grip) and Ladder Drill
  Interventions: Other: Drills

INTERVENTIONS:
Other: Plyometric Training — Ankle hops, jump squats, box jump, overhead medicine ball, plyometric push-up, rotational wall with 16x2 reps for week 1&2.
  Ankle hops, jump squats, box jump, overhead medicine ball, plyometric push-up, rotational wall with 10x3 reps for week 3&4.
  Ankle hops, jump squats, box jump, depth jump and alternate lunge jump, overhead medicine ball, plyometric push-up, rotational wall with 8x3 reps for week 5&6
  Arms: Plyometric Training
Other: Drills — Fast bowling drills (hitting a target, football throw, fast bowler grip) and Ladder Drill
  Arms: Drills

SUMMARY:
The sport of cricket calls for a high level of physical fitness and mastery of skills. Cricket players, especially fast bowlers, must have the skills to maintain consistency in their pace and accuracy while bowling helps them prevent batsmen from settling into their innings and helps bowlers succeed in getting wickets. Fast bowlers, being some of the most influential players on the cricket field, must undergo specific trainings. Sports-specific Drills and Plyometric training are two important types of training that help athletes in their particular sports.

DETAILED DESCRIPTION:
Randomized Clinical Trial (RCT) will be conducted to compare the effect of plyometric trainings versus bowling drills on speed and agility among fast bowlers. A sample size of 22 club level fast bowlers will be taken through Non-Probability Convenience Sampling Technique. One group of 11 participants will perform Plyometric training and other group of 11 participants will perform Bowling Drills and Ladder drill. Both groups will perform their respective trainings for 6 weeks with 3 sessions per week. Before and after completion of the respective training, speed, agility will be assessed through 30m sprint test, run-a-three test, illinois test, t-test respectively and bowling speed will be measured using a stopwatch to calculate the time required for the ball to reach a batsman and within 22 yards of the pitch. Data will be analyzed by using SPSS for windows version 25.

ELIGIBILITY:
Inclusion Criteria:

* Only male fast bowler will be recruited to the study.
* Athletes must have been practicing fast bowling for at least one year at the club level.
* Athletes must have been between the ages of 20-35.

Exclusion Criteria:

* Athletes who will have any systemic disease which can hinder the trainings.
* Athletes who would not commit to full participation in the study's training regimes.
* Athletes who have received surgery in the three years prior to the study or undergone rehabilitation within the past year.
* Athletes currently engaged in plyometric training as this may confound the study

Ages: 20 Years to 35 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Estimated)
Dates: Start 2023-03-25 (Actual); Primary Completion 2023-09-15 (Estimated); Study Completion 2023-10-22 (Estimated)

PRIMARY OUTCOMES:
T Test | 6 weeks
  The T-test is a measure of four-directional agility and body control. It measures the ability to change direction rapidly while maintaining balance without loss of speed. To perform the Agility T-Test a client is asked to run from the start point 10 meters forward to point one, sidestep to point two before sidestepping to point three, side stepping back to point one and then running back to the finish. The process is then repeated side stepping in the other direction first.
Run A Three Test | 6 weeks
  The Run-a-Three Test is a cricket fitness test that assesses both speed and agility in a very specific cricket situation. The run-a-three involves sprinting over the actual pitch distance three times, carrying a bat and incorporating two 180 degree turns. This test not only assesses speed, but also technique on the turn and running the bat in at the end.
Illinois Agility Test | 6 weeks
  The Illinois agility test is a fitness test designed to test one's sport agility. In which Participants should lie on their front (head to the start line) and hands by their shoulders. On the 'Go' command the stopwatch is started, and the athlete gets up as quickly as possible and runs forwards 10 meters to run around a cone, then back 10 meters, then runs up and back through a slalom course of four cones. Finally, the athlete runs another 10 meters up and back past the finishing cone, at which the timing is stopped.
30m Sprint Test | 6 weeks
  The 30m sprint test is to determine speed and acceleration. The test involves running a single maximum sprint over 30 meters, with the time recorded. Start from a stationary position, with one foot in front of the other. The tester provides hints for maximizing speed (such as keeping low, driving hard with the arms and legs) and encourage athletes to continue running hard through the finish line. Two trials are allowed, and the best time is recorded to the nearest 2 decimal places.
Bowling Speed Measure | 6 weeks
  It can be measured your bowling speed by using a stopwatch to calculate the time required for the ball to reach a batsman and within 22 yards of the pitch. Then, divide the distance by time and convert miles per hour or miles per hour.

CONTACTS AND LOCATIONS:
Overall Officials: Amna Shahid, t-DPT, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Raiwind Campus, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No